CLINICAL TRIAL: NCT06367335
Title: Characteristics and Predictors of Chemotherapy-induced Liver Injury in Advanced Breast Cancer Patients Treated With Cyclin-dependent Kinase Inhibitors CDK4/6
Brief Title: Characteristics and Predictors of Liver Injury in Cyclin-dependent Kinase Inhibitors 4/6 (CDK4/6)-Treated Patients With Advanced Breast Cancer
Acronym: ETIC
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Antonio Ciaccio, Principal Investigator, University of Milano Bicocca
Other Study IDs: ETIC
Record Dates: First submitted 2022-10-20; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: DILI
MeSH Terms: interventions — ribociclib; palbociclib; abemaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ribociclib, palbociclib, abemaciclib — evaluate the presence of predictors useful to predict the development of DILI during treatment with CKI

SUMMARY:
The main objective of the study is to evaluate the presence of predictors (single characteristics at the baseline and / or a combination of two or more parameters) useful for predicting the development of Drug-Induced liver Injury (DILI) during treatment with cyclin-dependent kinase inhibitors (CKI) with the possibility of obtaining a pre-treatment prognostic score that can assist the clinician in pre-therapy decision making.

DETAILED DESCRIPTION:
Drug Induced Liver Injury (DILI) is a rare liver disease that occurs as a reaction to exposure to drugs, herbal products and dietary supplements. Its onset is due to the interaction of several risk factors, associated with causative agent, host and environment. DILI is usually detected by an increase in liver enzymes with or without symptoms of liver disease1. It can occur with a variety of manifestations such as cholestasis, chronic hepatitis, steatosis, veno-occlusive disease and also neoplasm. According to last European Association for the Study of the Liver (EASL) guidelines, DILI should be suspected when one of the following thresholds is met, even in the absence of symptoms: alanine transferase (ALT) ≥ 5 times upper limit of normal (ULN), alkaline phosphatase (ALP) ≥ 2 ULN (particularly with accompanying elevations in concentrations of gamma-glutamyl transferase (GGT) in the absence of known bone pathology driving the rise in ALP level), total bilirubin concentration > 2 ULN associated with ALT ≥3 ULN. However, a stepwise clinical and laboratory approach is recommended to make the diagnosis of DILI.

The Roussel Uclaf Causality Assessment Method (RUCAM) scale has been demonstrated to be a valuable tool for assessing the possible causality of liver damage with the suspected drug. Liver biopsy should be performed only if discontinuation of the suspected culprit drug is not followed by improvement of liver damage after a reasonable observation period, or when autoimmune hepatitis (AIH) is suspected.

There are two types of DILI: the intrinsic direct form, which is dose-related and occurs early after agent exposure (hours or days), and the idiosyncratic indirect form, which is due to interactions between environment and host factors, and is not related to a threshold dose, with a longer latency period (a few days to several months). The incidence of this latter form is difficult to assess2 and is the one most observed during treatment with chemotherapy drugs.

There is mounting evidence of idiosyncratic DILI in patients with metastatic breast cancer (MBC) undergoing therapy with cyclin dependent kinases 4/6 (CDK4/6) inhibitors. Currently three CDK4/6 inhibitors have been approved for the treatment of MBC (palbociclib, ribociclib, and abemaciclib) and ribociclib has been reported to determine liver injury more frequently than the others.

Several randomized clinical trials have shown that these drugs improve both progression-free survival (PFS) and overall survival (OS) in Hormone receptor-positive (HR+)/human epidermal growth factor receptor 2-negative (HER2-) MBC with an acceptable toxicity profile. Recent reports have highlighted the distinct roles and occasional divergences between randomized controlled trials (RCTs) and population-based observational research, in general. The RCT rests on excellent internal validity, which is based on the randomization to ensure that the only difference between two treatment arms is their exposure to the treatment of interest. Given the differences between patients recruited to trials and those seen in routine practice, increased toxicity might be expected when the results of RCTs are applied to routine practice. Population-based studies can provide information about toxicity associated with treatment. With respect to the topic of our interest, although the incidence of adverse events seems comparable with that reported in RCTs, a higher incidence of treatment discontinuation with possible implications on treatment efficacy has been reported.

According to the experience of our Centre since the introduction of CDK4/6 inhibitors into clinical practice (unpublished data), toxicity of these drugs is apparently more frequent and severe than reported in previous publications, mainly registration trials, and, most importantly, produces a significant impact on the management of the treated patients, with a number of them needing temporary suspension, reintroduction at lower dose and even definitive withdrawal, without mention the burden of extra examinations prescribed and the concerns for the patient and her/his family. The weight of such treatment derailment on hard clinical outcomes has not been assessed yet, but it is certainly a potential cause of switching to less effective options.

ELIGIBILITY:
Inclusion Criteria:

* All patients with advanced breast cancer (Stage IV) consecutively evaluated at the Oncology Unit of our institution and who have received at least one dose of cyclin-dependent kinase inhibitors CDK4/6 (palbociclib, ribociclib, abemaciclib) since the European Union (EU) approval date (2016, 2017, 2018) and who have been followed-up for at least three months after the administration of the last dose of drug;
* Subjects willing to participate at the study data collection and aged at least 18.

Exclusion Criteria:

* Subjects with hepatocellular carcinoma (HCC).
* Subjects with chronic active hepatitis of any cause AND/OR cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by advanced breast cancer who are treated with regimens that include a cyclin-dependent kinase inhibitor (CKI).
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of DILI | 12 months
  Incidence of liver toxicity emerging on treatment, and defined according to EASL definition of drug-induced liver injury (DILI)

SECONDARY OUTCOMES:
withdrawal of therapy | 12 months
  Proportion of patients who had to stop antineoplastic therapy due to liver injury of any grade.
delayed reprise of antineoplastic therapy | 12 months
  Time interval of therapy missed for liver toxicity issues, in days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milano-Bicocca,, Monza, Italy

IPD SHARING:
Plan to Share IPD: No